CLINICAL TRIAL: NCT02075190
Title: Trial of a Nationwide Cognitive-Affective Remediation Training Intervention in Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Gyurak is no longer doing and ended her NARSAD early.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amit Etkin, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 28625
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cognitive-affective Exercises; Engaging Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Participants randomized to receive remediation training intervention delivered online (60 days of online training)
  Interventions: Other: Therapeutic Computerized intervention
- Control Group (Active Comparator): Participants randomized to receive online gaming intervention (60 days of online play)
  Interventions: Other: Nontherapeutic computerized intervention

INTERVENTIONS:
Other: Therapeutic Computerized intervention — Remediation training intervention
  Arms: Treatment Group
Other: Nontherapeutic computerized intervention — Online gaming intervention
  Arms: Control Group

SUMMARY:
The objective is to examine the efficacy of computerized interventions for increasing well-being and cognitive functioning. The study will seek to validate emerging online delivery methods of psychiatric assessment and treatment. This will allow us to test the efficacy of this intervention in a larger and more geographically broad sample than is possible through traditional recruitment and treatment, and to do so in a highly cost-effective manner.

ELIGIBILITY:
Inclusion Criteria:

* computer and broadband internet access
* 18 years of age
* Elevated anxiety and depression
* Native English speaker

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 1 month
  Behavioral measure of executive functions

SECONDARY OUTCOMES:
Self-report mood and anxiety symptoms | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anett Gyurak, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States